CLINICAL TRIAL: NCT01424813
Title: A 12-week Comparison of the Efficacy and Safety of Albuterol Spiromax® Versus Placebo in Subjects 12 Years and Older With Persistent Asthma
Brief Title: A 12-week Study to Compare the Efficacy and Safety of Albuterol Spiromax® Versus a Placebo in People 12 Years and Older With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-301
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Results first posted 2015-05-20 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
Keywords: Asthma; dry powder inhaler; short-acting beta2-agonist; SABA; bronchoconstriction; bronchodilation; bronchodilator; metered dose inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo MDPI (Placebo Comparator): Placebo multi-dose dry powder inhaler (MDPI) administered as 2 inhalations four times a day for 12 weeks.
  Interventions: Drug: Placebo MDPI
- Albuterol MDPI (Experimental): Albuterol multi-dose dry powder inhaler (MDPI) at a dose of 720 micrograms per day administered as 2 inhalations of 90 mcg /inhalation four times a day for 12 weeks.
  Interventions: Drug: Albuterol MDPI

INTERVENTIONS:
Drug: Placebo MDPI — Placebo MDPI administered as 2 inhalations 4 times a day (QID) (at approximately 7:00 AM, 12 noon, 5:00 PM, and bedtime) for 12 weeks.
  Other Names: Placebo Spiromax®
  Arms: Placebo MDPI
Drug: Albuterol MDPI — Albuterol MDPI administered as 2 inhalations 4 times a day (QID) (at approximately 7:00 AM, 12 noon, 5:00 PM, and bedtime) for 12 weeks.
  Other Names: ProAir® RespiClick, Albuterol Spiromax®
  Arms: Albuterol MDPI

SUMMARY:
The study will measure the change in lung function in subjects with asthma after inhaling from either of two inhalers: Albuterol Spiromax® or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent
* General good health
* Persistent asthma, with an FEV1 50-80% predicted.
* Ability to perform spirometry in an acceptable manner as per protocol guidelines.
* Ability to perform PEFR with a handheld peak flow meter.
* Demonstration of reversible bronchoconstriction as verified by a 15% or greater increase from baseline FEV1.
* Taking inhaled corticosteroids at a stable dose for at least 4 weeks prior to the Screening Visit.
* Non-smokers.
* Capable of understanding the requirements, risks, and benefits of study participation.
* Other inclusion criteria apply.

Exclusion Criteria:

* Participation in any investigational drug trial within the 30 days preceding the Screening Visit (SV).
* A known hypersensitivity to albuterol or any of the excipients in the formulations.
* History of severe milk protein allergy.
* History of a respiratory infection or disorder that has not resolved within the 2 weeks preceding the Screening Visit (SV).
* Currently requires treatment with β2-adrenergic receptor antagonists or non-selective β-receptor blocking agents.
* History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation.
* Any asthma exacerbation requiring oral corticosteroids within 3 months of the Screening Visit (SV). A subject must not have had any hospitalization for asthma within 6 months prior to the Screening Visit (SV).
* Historical or current evidence of any clinically significant non-asthmatic acute or chronic condition including.
* Other exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Leader, Study Director — Teva Respiratory R&D
Locations (38):
- United States (38):
  - Teva Investigational Site 10077, Birmingham, Alabama
  - Teva Investigational Site 10079, Phoenix, Arizona
  - Teva Investigational Site 10569, Costa Mesa, California
  - Teva Investigational Site 10053, Fountain Valley, California
  - Teva Investigational Site 10065, Huntington Beach, California
  - Teva Investigational Site 10572, Huntington Beach, California
  - Teva Investigational Site 10075, Los Angeles, California
  - Teva Investigational Site 10061, Roseville, California
  - Teva Investigational Site 10066, San Diego, California
  - Teva Investigational Site 10068, Denver, Colorado
  - Teva Investigational Site 10069, Denver, Colorado
  - Teva Investigational Site 10058, Miami, Florida
  - Teva Investigational Site 10060, Miami, Florida
  - Teva Investigational Site 10064, Ormond Beach, Florida
  - Teva Investigational Site 10071, Savannah, Georgia
  - Teva Investigational Site 10073, Wichita, Kansas
  - Teva Investigational Site 10070, Owensboro, Kentucky
  - Teva Investigational Site 10063, Bethesda, Maryland
  - Teva Investigational Site 10571, Gaithersburg, Maryland
  - Teva Investigational Site 10067, Wheaton, Maryland
  - Teva Investigational Site 10072, St Louis, Missouri
  - Teva Investigational Site 10050, Missoula, Montana
  - Teva Investigational Site 10057, Raleigh, North Carolina
  - Teva Investigational Site 10051, Cincinnati, Ohio
  - Teva Investigational Site 10078, Sylvania, Ohio
  - Teva Investigational Site 10054, Oklahoma City, Oklahoma
  - Teva Investigational Site 10568, Oklahoma City, Oklahoma
  - Teva Investigational Site 10055, Tulsa, Oklahoma
  - Teva Investigational Site 10056, Medford, Oregon
  - Teva Investigational Site 10076, Medford, Oregon
  - Teva Investigational Site 10684, Charleston, South Carolina
  - Teva Investigational Site 10570, Spartanburg, South Carolina
  - Teva Investigational Site 10049, Live Oak, Texas
  - Teva Investigational Site 10052, San Antonio, Texas
  - Teva Investigational Site 10685, Waco, Texas
  - Teva Investigational Site 10059, Fairfax, Virginia
  - Teva Investigational Site 10074, Puyallup, Washington
  - Teva Investigational Site 10062, Tacoma, Washington

REFERENCES:
- [Derived] Raphael G, Taveras H, Iverson H, O'Brien C, Miller D. Twelve- and 52-week safety of albuterol multidose dry powder inhaler in patients with persistent asthma. J Asthma. 2016;53(2):187-93. doi: 10.3109/02770903.2015.1070862. Epub 2015 Sep 15. PMID 26369589

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 384 patients screened; 180 patients were excluded on the basis of inclusion criteria, 4 due to exclusion criteria, 21 patients withdrew consent, 1 patient was lost to follow-up before the baseline visit, 6 patients had other reasons, and 14 patients failed to meet randomization criteria at the end of the run-in period.
Period: Overall Study
Arm/Group | Placebo MDPI | Albuterol MDPI
Started | 79 | 79
Treated | 79 (Safety set and full analysis set) | 78 (Safety set and full analysis set)
Completed | 74 | 77
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo MDPI | Albuterol MDPI | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (16.84) | 37.3 (16.89) | 38.8 (16.88)
Age, Customized [Number; unit: participants]
  12-17 years | 14 | 16 | 30
  18-64 years | 63 | 60 | 123
  65+ years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 44 | 91
  Male | 32 | 35 | 67
Race/Ethnicity, Customized [Number; unit: participants]
  White | 59 | 55 | 114
  Black | 18 | 21 | 39
  Asian | 2 | 0 | 2
  American Indian or Alaskan Native | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0
  Other | 0 | 3 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 76 | 73 | 149
Weight [Mean (Standard Deviation); unit: kg] | 82.4 (21.34) | 83.4 (24.20) | 82.9 (22.75)
Height [Mean (Standard Deviation); unit: cm] | 169.5 (9.47) | 168.9 (9.27) | 169.2 (9.35)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (6.92) | 29.2 (8.22) | 28.9 (7.58)

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) Over the 12-week Treatment Period
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. It represents the weighted average (by the trapezoidal rule) of FEV1 AUC 0-6 measures adjusted for the baseline measure (i.e., change from baseline at each timepoint) recorded on days 1, 8 and 85 of the treatment period. The baseline for each study day was the average of the 2 pre-dose FEV1 measurements on that study day.
  FEV1 was measured using spirometry. Spirometry assessments were obtained predose at -30 ± 5, and - 5 minutes, then post dose at 5 ± 2, 15 ± 5, 30 ± 5, 45 ± 5 minutes, and at 1hr ± 5 min, 2hr ± 5 min, 3hr ± 5 min, 4hr ± 5 min, 5hr ± 5 min, and 6hr ± 5 min.
Time Frame: Day 1, Day 8 and Day 85
Population: Full analysis set which includes all participants in the intent-to-treat (ITT) population who received at least 1 dose of study medication and had at least 1 post-baseline assessment.
Measure: Mean (Standard Error); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 79 | 78
L*hr | 0.28 (0.091) | 1.11 (0.092)
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed-model repeated-measures (MMRM) — Significance at the 0.05 level; Fixed effects- pooled center, treatment group, study day, and study day by drug interaction, with baseline measured at each study day as covariate; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.57 to 1.08], Standard Error of Mean 0.128

2. Secondary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) on Day 1
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. The baseline was the average of the 2 pre-dose FEV1 measurements on that study day. The baseline-adjustment refers to change from baseline at each post dose timepoint recorded on Day 1.
  FEV1 was measured using spirometry. Spirometry assessments were obtained predose at -30 ± 5, and - 5 minutes, then post dose at 5 ± 2, 15 ± 5, 30 ± 5, 45 ± 5 minutes, and at 1hr ± 5 min, 2hr ± 5 min, 3hr ± 5 min, 4hr ± 5 min, 5hr ± 5 min, and 6hr ± 5 min.
Time Frame: Day 1
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 79 | 78
L*hr | 0.52 [0.24 to 0.79] | 1.58 [1.30 to 1.87]
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures (MMRM) — To adjust for multiplicity, so that the overall alpha level for all tests was controlled at the 0.05 level, tests were done sequentially [day 1, then day 8, then day 85] and terminated if individual results were not significant at the 0.05 level; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.07, 95% CI 2-sided [0.68 to 1.46], Standard Error of Mean 0.198

3. Other Pre Specified Outcome: Percent Change From Baseline in FEV1 AUC 0-6 Over the 12-week Treatment Period
Time Frame: Day 1, Day 8, Day 85
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Percent Change From Baseline in FEV1 AUC 0-6
Time Frame: Day 1
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Percent Change From Baseline in FEV1 AUC
Time Frame: Day 8
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percent Change From Baseline in FEV1 AUC
Time Frame: Day 85
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Maximum Percent Change From Baseline in FEV1 Within 2 Hours Post Dose Over the 12-week Treatment Period
Time Frame: Day 1, Day 8, Day 85
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Maximum Percent Change From Baseline in FEV1 Within 2 Hours Post Dose on Day 1
Time Frame: Day 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Maximum Percent Change From Baseline in FEV1 Within 2 Hours Post Dose on Day 8
Time Frame: Day 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Maximum Percent Change From Baseline in FEV1 Within 2 Hours Post Dose on Day 85
Time Frame: Day 85
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Time to Onset of Effect (Change in FEV1 of 12% From Baseline Within 30 Minutes Postdose)
Time Frame: Day 1, Day 8, Day 85
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Duration of Response Measured From the Time Post-dosing to the First Time After the Response Onset (Increase ≥12% Above Baseline) When the FEV1 Decreases to Less Than 12% Above Baseline (Within 6 Hours After Dosing) for Those Who Responded in 30 Minutes
Time Frame: Day 1, Day 8, Day 85
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time to Onset of Effect (Change in FEV1 of 15% From Baseline Within 30 Minutes Postdose)for Those Who Responded in 30 Minutes
Time Frame: Day 1, Day 8, Day 85
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Duration of Response on Days 1, 8 and 85
Description: Duration of response measured from the time post-dosing to the first time after the response onset (increase ≥15% above baseline) when the FEV1 decreases to less than 15% above baseline (within 6 hours after dosing) for those who responded within 30 minutes
Time Frame: Day 1, Day 8, Day 85
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Percent of Symptom Free Days on the Patient Diary
Time Frame: Treatment days 1 through 85
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Percent of Rescue Medication Free Days in the Patient Diary
Time Frame: Treatment days 1 through 85
Reporting Status: Not Posted

17. Secondary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) on Day 8
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. The baseline was the average of the 2 pre-dose FEV1 measurements on that study day. The baseline-adjustment refers to change from baseline at each post dose timepoint recorded on Day 8.
  FEV1 was measured using spirometry. Spirometry assessments were obtained predose at -30 ± 5, and - 5 minutes, then post dose at 5 ± 2, 15 ± 5, 30 ± 5, 45 ± 5 minutes, and at 1hr ± 5 min, 2hr ± 5 min, 3hr ± 5 min, 4hr ± 5 min, 5hr ± 5 min, and 6hr ± 5 min.
Time Frame: Day 8
Population: Full analysis set of participants with data at the time point
Measure: Mean (95% Confidence Interval); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 78 | 78
L*hr | 0.26 [0.03 to 0.49] | 0.99 [0.76 to 1.22]
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [0.41 to 1.06], Standard Error of Mean 0.164

18. Secondary Outcome: Baseline-adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC 0-6) on Day 85
Description: FEV1 AUC 0-6 is the area under the effect-time curve from time 0 (pre-dose) up to 6 hours post-dose. The baseline was the average of the 2 pre-dose FEV1 measurements on that study day. The baseline-adjustment refers to change from baseline at each post dose timepoint recorded on Day 85.
  FEV1 was measured using spirometry. Spirometry assessments were obtained predose at -30 ± 5, and - 5 minutes, then post dose at 5 ± 2, 15 ± 5, 30 ± 5, 45 ± 5 minutes, and at 1hr ± 5 min, 2hr ± 5 min, 3hr ± 5 min, 4hr ± 5 min, 5hr ± 5 min, and 6hr ± 5 min.
Time Frame: Day 85
Population: Full analysis set of participants with data at the time point
Measure: Mean (95% Confidence Interval); unit: L*hr
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 77 | 77
L*hr | 0.06 [-0.15 to 0.28] | 0.74 [0.53 to 0.96]
Statistical Analysis 1: Comparison: Placebo MDPI vs Albuterol MDPI; Test type: Superiority or Other; p < 0.0001, mixed model repeated measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [0.38 to 0.99], Standard Error of Mean 0.154

19. Secondary Outcome: Participants With Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Day 92
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 79 | 78
participants
  Any adverse event | 25 | 22
  Severe adverse events | 1 | 1
  Treatment-related AE | 1 | 1
  Deaths | 0 | 0
  Other serious AEs | 0 | 0
  Withdrawn from study due to AEs | 0 | 0

20. Secondary Outcome: Physical Examination Findings Shifts From Baseline to Endpoint by Treatment Group
Description: Physical exam was recorded as normal or abnormal based on physician assessment. Format for results is: Test Baseline/Endpoint HEENT = head, eyes, ears, nose, throat
Time Frame: Day 1 (Baseline), Day 85
Population: Safety population. Only participants with both baseline and endpoint physical examination findings are summarized. Two placebo participants were missing endpoint physical examinations.
Measure: Number; unit: participants
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 77 | 78
participants
  General appearance Normal/Normal | 76 | 76
  General appearance Normal/Abnormal | 0 | 0
  General appearance Abnormal/Normal | 1 | 1
  General appearance Abnormal/Abnormal | 0 | 1
  HEENT Normal/Normal | 46 | 50
  HEENT Normal/Abnormal | 12 | 5
  HEENT Abnormal/Normal | 11 | 12
  HEENT Abnormal/Abnormal | 8 | 11
  Chest and Lungs Normal/Normal | 66 | 67
  Chest and Lungs Normal/Abnormal | 8 | 4
  Chest and Lungs Abnormal/Normal | 2 | 7
  Chest and Lungs Abnormal/abnormal | 1 | 0
  Heart Normal/Normal | 76 | 77
  Heart Normal/Abnormal | 0 | 0
  Heart Abnormal/Normal | 1 | 1
  Heart Abnormal/Abnormal | 0 | 0
  Abdomen Normal/Normal | 75 | 77
  Abdomen Normal/Abnormal | 1 | 0
  Abdomen Abnormal/Normal | 0 | 1
  Abdomen Abnormal/Abnormal | 1 | 0
  Musculoskeletal Normal/Normal | 74 | 76
  Musculoskeletal Normal/Abnormal | 0 | 1
  Musculoskeletal Abnormal/Normal | 3 | 1
  Musculoskeletal Abnormal/Abnormal | 0 | 0
  Skin Normal/Normal | 75 | 73
  Skin Normal/Abnormal | 0 | 1
  Skin Abnormal/Normal | 2 | 4
  Skin Abnormal/Abnormal | 0 | 0
  Lymph nodes Normal/Normal | 77 | 78
  Lymph nodes Normal/Abnormal | 0 | 0
  Lymph nodes Abnormal/Normal | 0 | 0
  Lymph nodes Abnormal/Abnormal | 0 | 0
  Neurological Normal/Normal | 76 | 78
  Neurological Normal/Abnormal | 1 | 0
  Neurological Abnormal/Normal | 0 | 0
  Neurological Abnormal/Abnormal | 0 | 0

21. Secondary Outcome: Participants With Clinically Significant Vital Sign Assessments
Description: For both standard and serial vital signs, participants were seated for at least 5 minutes before vital signs were assessed. Heart rate was obtained prior to the blood pressure measurement. Serial heart rate and blood pressure were conducted in the sitting position prior to the spirometry assessment; baseline measures were taken pre-dose at -30 ± 5 and -5 minutes on Day 1. Day 85 serial vital sign measures were taken in the sitting position prior to spirometry assessments pre-dose at -30 ± 5 and -5 minutes, then post-dose at 30 (±5) minutes, 1hr (± 10 min), 2hr (± 10 min), 3hr (± 10 min), 4hr (± 10 min), 5hr (± 10 min) and 6 hr (± 10 min).
  Serial heart rate and blood pressure measurements that were elevated to the following criteria were considered clinically significant:
  Systolic blood pressure: > 160 beats/minute Diastolic blood pressure: >100 beats/minute Heart rate: >120 beats/minute
Time Frame: Day 8, Day 85
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Placebo MDPI | Albuterol MDPI
Number analyzed (Participants) | 79 | 78
participants
  Systolic blood pressure - high | 3 | 0
  Diastolic blood pressure - high | 3 | 1
  Heart rate - high | 0 | 1

22. Other Pre Specified Outcome: Morning Peak Expiratory Flow Reading Reported on Patient Diary
Time Frame: Treatment days 1 through 85
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 1 to Day 92
Arm/Group | Albuterol MDPI | Placebo MDPI
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/79
Other Adverse Events (participants affected / at risk) | 6/78 | 9/79
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol MDPI (N=78) | Placebo MDPI (N=79)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 3 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.